CLINICAL TRIAL: NCT01653600
Title: Efficacy of Self-Expanding Nitinol S.M.A.R.T CONTROLTM Stent Versus Life Stent For The Atherosclerotic Femoro-Popliteal Arterial Disease : Prospective, Multicenter, Randomized, Controlled Trial (SENS-FP-2 Trial)
Brief Title: Efficacy of Self-Expanding Nitinol S.M.A.R.T CONTROL Stent Versus Life Stent For The Atherosclerotic Femoro-Popliteal Arterial Disease
Acronym: SENS-FP-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Associate professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENS-FP-2-LifeStent Arm
Record Dates: First submitted 2012-04-09; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis
Keywords: peripheral arterial disease; atherosclerosis; nitinol; stents
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LifeStent (Experimental): same to SMART CONTROL Stent
  Interventions: Device: LifeStent
- SMART CONTROL Stent (Active Comparator): study design is 2x2 randomization design. First, before randomization, stratification will be performed according to lesion length 15cm criteria at web-based computerized program. Patients will be randomized in a 1:1 manner according to different two (SMART versus LifeStent) stents. And then, patients received aspirin and clopidogrel during one month. After one month from index procedure, clopidogrel will be stopped and changed into cilostazol. Patients were randomized to receive cilostazol 100mg bid either 11 month duration or 5 month duration in separate groups of SMART stent group and LifeStent group. Randomization procedure will be performed using a web-based program
  Interventions: Device: S.M.A.R.T CONTROL Stent

INTERVENTIONS:
Device: S.M.A.R.T CONTROL Stent — Provisional stenting should be performed; the case that optimal ballooning response is not obtained (sub-optimal balloon response) should be enrolled. The procedure is usually done, as follows; After the guidewire is passed through the target lesion, predilation of the target lesion with an optimally sized balloon will be performed prior to stent implantation. Recommended, minimal balloon dilation time is 120 seconds. The sub-optimal balloon response is defined as a residual pressure gradient of >15 mmHg, residual stenosis of >30%, and flow-limiting dissection.
  Arms: SMART CONTROL Stent
Device: LifeStent — same to SMART STENT
  Arms: LifeStent

SUMMARY:
The nitinol stent has proven superior primary patency than balloon angioplasty in superficial femoral artery lesions. Recent stent design improvements focus on decreasing stent fracture rates which can negatively impact patency rates by rearranging strut alignment. In the literature, however, prospective, randomized, controlled, clinical trial for comparison of stent fracture and primary patency between different nitinol stents has never been performed except one study; SMART versus Luminexx stent named SuperSL trial. LifeStent is similar to S.M.A.R.T. stent in the design consisted of the peak-to-valley connected with S-shaped bridge but is different in lesser bridge (4 bridge vs. 6 bridge), large cell size on stent ends, and larger cell size than S.M.A.R.T. On the other hand, Recent meta-analysis has shown that the efficaty of cilostazol in the atherosclerotic femoropopliteal lesion was proven. However, still specific data regarding a variety of antiplatelet regimen in implanted femoropopliteal lesion are limited. Upto date, in the literature, never has never been performed the clinical trial for optimal duration of cilostazol use in the patient undergone stent implantation for femoropopliteal lesion. Thus, The purpose of our study is to examine and compare Primary patency and stent fracture between different two-nitinol stents (S.M.A.R.T. CONTROL versus Lifestent) in femoropopliteal arterial lesion and to examine and compare the optimal duration of cilostazol use.

DETAILED DESCRIPTION:
Five randomized, controlled trials failed to demonstrate any benefit of a stainless-steel stent over angioplasty alone. The nitinol stent has proven superior primary patency than balloon angioplasty in superficial femoral artery lesions. Recent stent design improvements focus on decreasing stent fracture rates which can negatively impact patency rates by rearranging strut alignment. In vitro, Stefan et al. reported difference in stent design might play a major role in the appearance of stent strut fracture related to restenosis and reocclusion. Also, several retrospective or registry clinical studies reported stent fractures were associated with a higher risk of in-stent restenosis and reocclusion. In the literature, however, prospective, randomized, controlled, clinical trial for comparison of stent fracture and primary patency between different nitinol stents has never been performed except one study; SMART versus Luminexx stent named SuperSL trial (lesion length between 5-22 cm). Furthermore, in the Asian population, the study of this type have never been performed. LifeStent is similar to S.M.A.R.T. stent in the design consisted of the peak-to-valley connected with S-shaped bridge but is different in lesser bridge (4 bridge vs. 6 bridge), large cell size on stent ends, and larger cell size than S.M.A.R.T. On the other hand, 2011 ESC guideline recommended that dual antiplatelet therapy with aspirin and a thienopyridine for at least one month is recommended after infrainguinal bare-metal-stent implantation. Recent meta-analysis has shown that the efficaty of cilostazol in the atherosclerotic femoropopliteal lesion was proven. However, still specific data regarding a variety of antiplatelet regimen in implanted femoropopliteal lesion are limited. Upto date, in the literature, never has never been performed the clinical trial for optimal duration of cilostazol use in the patient undergone stent implantation for femoropopliteal lesion. Thus, The purpose of our study is to examine and compare Primary patency and stent fracture between different two-nitinol stents (S.M.A.R.T. CONTROL versus Lifestent) in femoropopliteal arterial lesion and to examine and compare the optimal duration of cilostazol use (6 month versus 12 month)

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria

  1. Age 20 years of older
  2. Symptomatic peripheral-artery disease with (Rutherford 2 - 6); moderate to severe claudication (Rutherford 2-3), chronic critical limb ischemia with pain while was at rest (Rutherford 4), or with ischemic ulcers (Rutherford 5-6)
  3. Patients with signed informed consent
* Anatomical criteria

  1. Target lesion length < 3 cm by angiographic estimation
  2. Stenosis of >50% or occlusive atherosclerotic lesion of the ipsilateral femoropopliteal artery
  3. Patent (≤50% stenosis) ipsilateral iliac artery or concomitantly treatable ipsilateral iliac lesions (≤30% residual stenosis),
  4. At least one patent (less than 50% stenosed) tibioperoneal run-off vessel.

Exclusion Criteria:

1. Disagree with written informed consent
2. Major bleeding history within prior 2 months
3. Known hypersensitivy or contraindication to any of the following medication: heparin, aspirin, clopidogrel or contrast agent
4. Acute limb ischemia
5. Previous bypass surgery or stenting of the ipsilateral femoropopliteal artery
6. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)
7. Patients that major amputation ("above the ankle" amputation) has been done, is planned or required
8. Patients with life expectancy <1 year due to comorbidity
9. end-staged renal failure on hemodialysis or peritoneal dialysis
10. Age > 85 years

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The rate of binary restenosis | one year
  binary restenosis is defined as the restenosis of at least 50 percent of the luminal diameter in the treated segment at 12 months after intervention, when determined by catheter angiography.

SECONDARY OUTCOMES:
stent fracture rate, clinical outcomes, angiographic outcomes, ankle-brachial index | 1 year
  1. Stent fracture rate
  2. Limb salvage free of above-the-ankle amputation
  3. Sustained clinical improvement rate
  4. Repeated target lesion revascularization rate
  5. Repeated target extremity revascularization rate
  6. Total re-occlusion rate
  7. Anigoraphic variables (Late loss, % restenosis)
  8. Ankle-brachial index
  9. The rate of major adverse cardiovascular events (MACE)
  10. The incidence of the stent geographic miss during stent deployment
  11. binary restenosis rate according to cilostazol use duration upto 12 month and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Woon Rha, MD, PhD, Principal Investigator — Cardiovascular Center, Korea University Guro Hospital, 80, Guro-dong, Guro-gu, Seoul, 152-703, Korea
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea